CLINICAL TRIAL: NCT02826668
Title: Pre-insertion Ultrasound Guidance for Labor Epidural Placement in the Lateral Position: A Randomized Controlled Trial of Image Reproducibility During Labor and Impact on Resident Learning Curve
Brief Title: Influence of Lumbar Ultrasound on Resident Learning Curve for Lateral Labor Epidural Placement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to loss of study staff and inability to recruit patients during COVID 19
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Michaela Kristina Farber, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2013P002510
Record Dates: First submitted 2016-06-26; First posted 2016-07-11 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Labor Epidural; Lumbar Ultrasound
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Baseline ultrasound only, with no markings placed. No ultrasound prior to epidural placement.
- Ultrasound (Experimental): Baseline and pre-puncture ultrasound with markings placed.
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — A baseline lumbar ultrasound in a standardized lateral position (by bed markings) will be performed with the midline and L3-L4 interspace marked, and estimated depth to the epidural space recorded. A second lateral lumbar ultrasound will be performed immediately prior to placement at the time of epidural request. The bed position will be standardized with lines drawn down the back, at the flexion of the knee, and heel of the foot. The sonographic measurements will include the midline, the L3-4 interspace, (both marked at the skin surface), and the measured depth to the ligamentum flavum (in centimeters).
  Arms: Ultrasound

SUMMARY:
The aim of this study is to evaluate the impact of lumbar spine ultrasound on the success rate and efficiency of labor epidural placement in the lateral position. The investigators hypothesize that ultrasound imaging of the lumbar spine of women in early labor will yield similar ultrasound results when done immediately prior to epidural placement. The investigators also hypothesize that the use of ultrasound with landmarks marked and depth to the epidural space estimated will facilitate epidural placement in terms of both efficiency (time required for placement) and efficacy of pain relief.

DETAILED DESCRIPTION:
Several studies have demonstrated a significant benefit in pre-procedural ultrasound for epidural placement by anesthesia residents, particularly when performed in the obese population. To the investigators knowledge, however, no studies have evaluated this teaching modality for the lumber epidural technique in the lateral position. Formalizing the educational process for this less frequently performed, highly technical and critical skill may have a profound impact on trainee learning curves, and may enhance the overall success and efficiency of epidural placement, quality of analgesia provided, and safety of the procedure.

ELIGIBILITY:
Pregnant Subjects

Inclusion Criteria:

* pregnant women
* 18 years or older
* in early labor (cervix dilated < 5 cm
* pain visual analog score (VAS) < 3, or both) requesting consultation by the anesthesia team for anticipated epidural pain relief.

Exclusion Criteria:

* absolute contraindications of neuraxial anesthesia including patient refusal
* uncorrected coagulopathy
* infection at the skin site of epidural placement
* increased intracranial pressure, or untreated hemodynamic instability.
* In addition, patients with a history of scoliosis or spine surgery
* body mass index (BMI) >40 kg/m2
* allergy to local anesthetic, or allergy to opioids will be excluded.

Anesthesiologists

Inclusion criteria:

* Anesthesia residents or fellows who are performing the epidural technique in pregnant subjects who agree to be part of the study.
* Anesthesia residents or fellows with prior experience in the lumbar epidural technique, defined as having placed 20 or greater lumbar epidurals during their residency and prior to enrollment.

Exclusion criteria:

* individuals who do not want to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-06; Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Depth to the epidural space (cm) from baseline ultrasound compared to pre-placement ultrasound. | From enrollment to time of epidural placement, approximately 5 hours
  Measured depth to the epidural space (cm) from baseline ultrasound compared to pre-placement ultrasound, measured with a 2-5 MHz curvilinear ultrasound probe at the lumbar spine, midline, at level L3-4.
Time required for epidural placement | From enrollment to time of epidural placement, approximately 5 hours
  Time required for placement (T0 = insertion of needle for subcutaneous lidocaine infusion prior to epidural needle placement). Tfinal = time at complete removal of Weiss epidural needle after catheter is threaded into the epidural space.
Need for assistance from additional anesthesiologist | From enrollment to time of epidural placement, approximately 5 hours
  Need for assistance from additional anesthesiologist
Number of attempts at epidural placement | From enrollment to time of epidural placement, approximately 5 hours
  defined as number of times the Weiss epidural needle enters the skin
Incidence of paresthesias | From enrollment to time of epidural placement, approximately 5 hours
  Paresthesia defined as pain with needle or catheter insertion
Labor pain at time of 30 minutes after placement is complete. | From enrollment to time of epidural placement, approximately 5 hours, plus 30 minutes.
  Labor pain rated on a visual analog scale (VAS)
Rate of epidural replacement for inadequate analgesia | From enrollment to time of epidural placement, approximately 5 hours
  Inadequate analgesia determined as VAS >3 despite catheter adjustment and/or epidural dose adjustment.
Rate of inadvertent dural puncture at the time of placement. | From enrollment to time of epidural placement, approximately 5 hours
  Defined as cerebrospinal fluid aspiration through needle or catheter.
Midline measurement from baseline ultrasound compared to pre-placement ultrasound. | From enrollment to time of epidural placement, approximately 5 hours
  Measured midline (anatomical marking) from baseline ultrasound compared to pre-placement ultrasound, measured with a 2-5 MHz curvilinear ultrasound probe at the lumbar spine, midline.
L3-L4 lumbar spine level measured from baseline ultrasound compared to pre-placement ultrasound. | From enrollment to time of epidural placement, approximately 5 hours
  Measured L3-L4 lumbar spine level from baseline ultrasound compared to pre-placement ultrasound, measured with a 2-5 MHz curvilinear ultrasound probe at the lumbar spine, paramedic.

CONTACTS AND LOCATIONS:
Overall Officials: Michaela K Farber, MD MS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mhyre JM, Greenfield ML, Tsen LC, Polley LS. A systematic review of randomized controlled trials that evaluate strategies to avoid epidural vein cannulation during obstetric epidural catheter placement. Anesth Analg. 2009 Apr;108(4):1232-42. doi: 10.1213/ane.0b013e318198f85e. PMID 19299793
- [Background] Harney D, Moran CA, Whitty R, Harte S, Geary M, Gardiner J. Influence of posture on the incidence of vein cannulation during epidural catheter placement. Eur J Anaesthesiol. 2005 Feb;22(2):103-6. doi: 10.1017/s0265021505000190. PMID 15816587
- [Background] Grau T, Bartusseck E, Conradi R, Martin E, Motsch J. Ultrasound imaging improves learning curves in obstetric epidural anesthesia: a preliminary study. Can J Anaesth. 2003 Dec;50(10):1047-50. doi: 10.1007/BF03018371. PMID 14656785
- [Background] Vallejo MC, Phelps AL, Singh S, Orebaugh SL, Sah N. Ultrasound decreases the failed labor epidural rate in resident trainees. Int J Obstet Anesth. 2010 Oct;19(4):373-8. doi: 10.1016/j.ijoa.2010.04.002. Epub 2010 Aug 8. PMID 20696564
- [Background] Balki M. Locating the epidural space in obstetric patients-ultrasound a useful tool: continuing professional development. Can J Anaesth. 2010 Dec;57(12):1111-26. doi: 10.1007/s12630-010-9397-y. Epub 2010 Nov 11. English, French. PMID 21063818
- [Background] Sahin T, Balaban O, Sahin L, Solak M, Toker K. A randomized controlled trial of preinsertion ultrasound guidance for spinal anaesthesia in pregnancy: outcomes among obese and lean parturients: ultrasound for spinal anesthesia in pregnancy. J Anesth. 2014 Jun;28(3):413-9. doi: 10.1007/s00540-013-1726-1. Epub 2013 Oct 20. PMID 24141882
- [Background] Carvalho JC. Ultrasound-facilitated epidurals and spinals in obstetrics. Anesthesiol Clin. 2008 Mar;26(1):145-58, vii-viii. doi: 10.1016/j.anclin.2007.11.007. PMID 18319185
- [Result] Grau T, Leipold RW, Fatehi S, Martin E, Motsch J. Real-time ultrasonic observation of combined spinal-epidural anaesthesia. Eur J Anaesthesiol. 2004 Jan;21(1):25-31. doi: 10.1017/s026502150400105x. PMID 14768920